CLINICAL TRIAL: NCT02196610
Title: Arterial Stiffness in Healthy Subjects and Patients With End-Stage- Renal Disease: A Feasibility Study
Brief Title: Feasibility Study of Arterial Stiffness in Hemodialysis Patients
Status: Terminated | Type: Observational
Why Stopped: Limited funds available to complete full recruitment. Enrolment achieved: 90%.
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital (Other); University of Ottawa (Other)
Responsible Party: Sponsor
Other Study IDs: 20140457
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-03

CONDITIONS: End-Stage Renal Disease
Keywords: End-Stage Renal Disease,; arterial or vascular stiffness,; hemodialysis,; Pulse wave velocity; Renal insufficiency,; tonometry
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HEALTHY SUBJECTS group: A group of 20 healthy staff volunteers identified from the Division of Nephrology, Dept. of Medicine and the Kidney Research Centre at the Ottawa Hospital Research Institute will be invited to participate. Measurements of arterial stiffness will be performed by Applanation tonometry. Healthy status will be defined by a self-reporting questionnaire obtained over the phone prior to enrolment and 2 subsequent non-invasive measurements of arterial blood pressure (BP) prior to testing. Subjects will be included if diastolic BP is ≤ 90 mm Hg and systolic BP ≤ 140 mm Hg on 2 consecutive measurements.
  Interventions: Other: Applanation tonometry
- END-STAGE RENAL DISEASE (ESRD) group: A group of 20 patients with stage 5 Chronic Kidney Disease (estimated glomerular filtration rate <15 ml/min/m2), who attend chronic hemodialysis treatments at The Ottawa Hospital (TOH) will be invited to participate. Measurements of arterial stiffness will be performed in this group by Applanation tonometry.
  Interventions: Other: Applanation tonometry

INTERVENTIONS:
Other: Applanation tonometry — Two consecutive sets of carotid-femoral Pulse Wave Velocity (PWV) measurements by Applanation tonometry with a time-interval of 1 week will be obtained (1 week ± 2 days). Two research assistants will each perform a carotid-femoral-PWV measurement at each time point with the testing order randomized.
  Other Names: carotid-femoral Pulse wave velocity (c-f-PWV)

SUMMARY:
People with kidney failure have a higher chance of getting disease in the blood vessels and this result in a decreased elasticity of the arteries of their body which make them very stiff or hard. It appears that stiffer arteries with a decreased elasticity increase the risk of stroke and heart disease. A novel way to know the stiffness of blood vessels is by a method called "applanation tonometry", which measures the "pulse wave velocity" of major blood vessels such as the aorta, carotid and femoral arteries. The purpose of our study is to determine if we can measure arterial stiffness reliably and accurately using this method in healthy people and in people with kidney failure receiving hemodialysis treatments at our centre. Also, we would like to know how stiff these arteries in healthy people are. If we demonstrate that the method is reliable and accurate in these 2 groups of participants at our centre, a future larger study is planned to determine if we can use measures of arterial stiffness to evaluate the risk of stroke and heart disease in people with kidney failure receiving hemodialysis. The research study will take place at the Ottawa Hospital-Riverside Campus.

DETAILED DESCRIPTION:
Background:

Cardiovascular (CV) disease is a major cause of morbidity and mortality in patients with end-stage renal disease (ESRD). Arterial stiffness measured by pulse-wave velocity (PWV) has been identified as an independent predictor of fatal CV events in these patients. Our long-term goal is to study the impact of interventions that decrease progressive arterial stiffness on CV mortality in ESRD patients. Thus, we postulate that measurements of PWV during these interventions will predict CV outcome. Before studying this relationship, establishing the feasibility of PWV measurements at our centre is necessary.

Objectives:

i) To demonstrate the reliability and accuracy of arterial PWV measurements in healthy subjects and patients with ESRD at our centre, ii) To assess subject satisfaction and level of discomfort associated with the testing procedure, iii) To characterize normative values for the PWV in our two subject groups, and iv) To determine the feasibility of recruitment of patients with ESRD, as a pre-requisite for a larger trial focused on CV outcomes.

Methods:

PWV will be measured consecutively by 2 research assistants in: a) a group of 20 healthy subjects; and b) a group of 20 patients with ESRD on chronic hemodialysis at The Ottawa Hospital. Two consecutive sets of PWV measurements with a time-interval of 1 week (± 2 days) will be obtained in the healthy and ESRD groups (pre-hemodialysis, between 2 consecutive mid-week hemodialysis sessions). To determine the impact of hemodialysis on PWV measures, in a sub-group of 10 ESRD subjects measurements will be taken before and after hemodialysis. The order of testing by the 2 assistants will be randomized.

ELIGIBILITY:
HEALTHY SUBJECT GROUP

Inclusion criteria:

* Age: >18 years
* Able to provide informed consent

Exclusion criteria

* History of cardiovascular disease and/or hypertension (blood pressure >140/90 mm Hg)
* History of diabetes mellitus
* History of liver or kidney disease, cancer and/or any lymphoproliferative disease
* Currently receiving medication for any medical condition or illness
* Body Mass Index (BMI) ≥ 30 Kg/m2
* Pregnancy
* Any condition that limits functional ability and precludes participation
* Current smoker (>15 cigarettes per day) in the last 6 months.
* Former smoker (> 20 cigarettes per day) who stopped smoking < 2 years ago.
* Excessive alcohol intake (men >14 drinks per week; women: > 9 drinks per week).
* Psychoactive or performance-enhancing drug abuse.

END-STAGE RENAL DISEASE (ESRD) GROUP

Inclusion Criteria:

* Adult patient (age: >18 years) with ESRD (estimated glomerular filtration rate: <15 ml/min/m2)
* Receiving hemodialysis treatments, with no expected renal recovery
* Having received regular in-Centre Hemodialysis at TOH for at least the past 3 weeks
* Able to provide informed consent.

Exclusion Criteria:

* Atrial fibrillation (as it frequently results in transient or persistent rapid heart rates and these changes overestimate aortic stiffness).
* Active cancer or history of cancer in the past 5 years.
* Pregnancy
* Any condition that limit the patient's ambulatory ability and preclude participation on this basis
* Mechanical, bioprosthetic heart valves or mechanical assisting devices (these conditions may change myocardial stiffness and the volumetric properties of the left ventricle leading to diastolic dysfunction and these physiologic changes may modify the waveforms of the cf- APWV).
* Pre-dialysis systolic blood pressure ≥ 200 mm Hg recorded in the last 6 dialysis treatments (2 weeks).
* Inability to measure blood pressure in at least one arm.
* Current smoker (>15 cigarettes per day) in the last 6 months [Daily cigarette consumption (>15 cigarettes per day) adjusted by age, education level and other confounders has been found to be independently associated with the risk of hypertension].

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HEALTHY SUBJECTS: 20 healthy staff volunteers.
  ESRD group: 20 patients with stage 5 CKD (estimated GFR <15 ml/min/m2), who attend chronic hemodialysis treatments at The Ottawa Hospital (TOH).
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Reliability of carotid-femoral Pulse Wave Velocity measurements | 1 week
  We will estimate the Pulse Wave Velocity differences and the intra-class correlation coefficient (ICC) between the 2 examinations (test-retest) recorded in the same subject 1 week apart. We will also estimate the examiner's reliability by the inter-rater agreement through the ICC and limits of agreement.

SECONDARY OUTCOMES:
Accuracy of the carotid-femoral Pulse Wave Velocity measurements | 1 week
  This will be estimated by calculating the mean, standard deviation and 95% confidence interval of the Pulse Wave Velocity differences between our healthy group and the age-adjusted mean values from a historical healthy control group
Subject satisfaction and procedure discomfort | 1 week
  This will be accomplished by surveying subjects at the end of the testing procedure using a Likert-type questionnaire
Recruitment Efficacy | 11 months
  We will assess the proportion of patients with End-Stage Renal disease (ESRD) who consented to the testing procedure relative to the number of eligible and screened participants

OTHER OUTCOMES:
Normative Pulse Wave Velocity Values | 11 months
  We will calculate the mean, standard deviation and 95% confidence interval of the pulse wave velocity values and Augmentation index in our defined populations.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Burns, MD, CM, Study Director — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital - Riverside campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] Moody WE, Edwards NC, Chue CD, Ferro CJ, Townend JN. Arterial disease in chronic kidney disease. Heart. 2013 Mar;99(6):365-72. doi: 10.1136/heartjnl-2012-302818. Epub 2012 Oct 31. PMID 23118349
- [Background] Vlachopoulos C, Aznaouridis K, Stefanadis C. Prediction of cardiovascular events and all-cause mortality with arterial stiffness: a systematic review and meta-analysis. J Am Coll Cardiol. 2010 Mar 30;55(13):1318-27. doi: 10.1016/j.jacc.2009.10.061. PMID 20338492
- [Background] Guerin AP, Blacher J, Pannier B, Marchais SJ, Safar ME, London GM. Impact of aortic stiffness attenuation on survival of patients in end-stage renal failure. Circulation. 2001 Feb 20;103(7):987-92. doi: 10.1161/01.cir.103.7.987. PMID 11181474
- [Background] Karras A, Haymann JP, Bozec E, Metzger M, Jacquot C, Maruani G, Houillier P, Froissart M, Stengel B, Guardiola P, Laurent S, Boutouyrie P, Briet M; Nephro Test Study Group. Large artery stiffening and remodeling are independently associated with all-cause mortality and cardiovascular events in chronic kidney disease. Hypertension. 2012 Dec;60(6):1451-7. doi: 10.1161/HYPERTENSIONAHA.112.197210. Epub 2012 Oct 22. PMID 23090769
- [Background] Pannier B, Guerin AP, Marchais SJ, Safar ME, London GM. Stiffness of capacitive and conduit arteries: prognostic significance for end-stage renal disease patients. Hypertension. 2005 Apr;45(4):592-6. doi: 10.1161/01.HYP.0000159190.71253.c3. Epub 2005 Mar 7. PMID 15753232
- [Background] Boutouyrie P, Fliser D, Goldsmith D, Covic A, Wiecek A, Ortiz A, Martinez-Castelao A, Lindholm B, Massy ZA, Suleymanlar G, Sicari R, Gargani L, Parati G, Mallamaci F, Zoccali C, London GM. Assessment of arterial stiffness for clinical and epidemiological studies: methodological considerations for validation and entry into the European Renal and Cardiovascular Medicine registry. Nephrol Dial Transplant. 2014 Feb;29(2):232-9. doi: 10.1093/ndt/gft309. Epub 2013 Sep 30. PMID 24084326
- [Background] Frimodt-Moller M, Nielsen AH, Kamper AL, Strandgaard S. Reproducibility of pulse-wave analysis and pulse-wave velocity determination in chronic kidney disease. Nephrol Dial Transplant. 2008 Feb;23(2):594-600. doi: 10.1093/ndt/gfm470. Epub 2007 Nov 7. PMID 17989106
- [Background] Reference Values for Arterial Stiffness' Collaboration. Determinants of pulse wave velocity in healthy people and in the presence of cardiovascular risk factors: 'establishing normal and reference values'. Eur Heart J. 2010 Oct;31(19):2338-50. doi: 10.1093/eurheartj/ehq165. Epub 2010 Jun 7. PMID 20530030
- [Background] Pan CR, Schmaderer C, Roos M, von Eynatten M, Sollinger D, Lutz J, Heemann U, Baumann M. Comparing aortic stiffness in kidney transplant recipients, hemodialysis patients, and patients with chronic renal failure. Clin Transplant. 2011 Jul-Aug;25(4):E463-8. doi: 10.1111/j.1399-0012.2011.01462.x. Epub 2011 Apr 26. PMID 21517999
- [Background] Giraudeau B, Mary JY. Planning a reproducibility study: how many subjects and how many replicates per subject for an expected width of the 95 per cent confidence interval of the intraclass correlation coefficient. Stat Med. 2001 Nov 15;20(21):3205-14. doi: 10.1002/sim.935. PMID 11746313
- [Background] Cavalcante JL, Lima JA, Redheuil A, Al-Mallah MH. Aortic stiffness: current understanding and future directions. J Am Coll Cardiol. 2011 Apr 5;57(14):1511-22. doi: 10.1016/j.jacc.2010.12.017. PMID 21453829
- [Derived] Rodriguez RA, Cronin V, Ramsay T, Zimmerman D, Ruzicka M, Burns KD. Reproducibility of carotid-femoral pulse wave velocity in end-stage renal disease patients: methodological considerations. Can J Kidney Health Dis. 2016 Apr 1;3:20. doi: 10.1186/s40697-016-0109-6. eCollection 2016. PMID 27042326